CLINICAL TRIAL: NCT03562520
Title: Toward Exercise as Medicine for Adolescents With Bipolar Disorder: A Feasibility Study
Brief Title: Toward Exercise as Medicine for Adolescents With Bipolar Disorder
Acronym: TEAM-BD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to the COVID-19 pandemic as no in-person study visits were permitted.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of British Columbia (Other); The Hospital for Sick Children (Other); Mood Disorders Association of Ontario (Unknown)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Senior Scientist, Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007-2018
Record Dates: First submitted 2018-04-23; First posted 2018-06-19 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
Keywords: Aerobic fitness; Aerobic exercise; Behavior change counseling
MeSH Terms: conditions — Bipolar Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with bipolar disorder (Experimental): Forty adolescents (aged 13-21) with BD (type I, II, or not otherwise specified/other specified and related disorder) will be enrolled in the behavior change counseling intervention.
  Interventions: Behavioral: Behavior change counseling

INTERVENTIONS:
Behavioral: Behavior change counseling — Core modules: 1 psychoeducation session at week 0; 4 behavior change counseling (BCC) sessions will occur at weeks 0, 4, 8, and 12; phone calls and/or texting sessions (weeks 1-3, 5-7, 9-11, and "booster" calls and/or texts on weeks 16 and 20) from therapists.
  Optional modules: Exercise coaching sessions; family involvement options will include participation in any aspect of the intervention; peer support options will include: group exercise classes on site, online Fitbit groups where adolescents can participate in competitions with each other and provide motivational support, and fitness support groups facilitated by registered social workers.

SUMMARY:
This study seeks to bridge the knowledge-to-action gap regarding "exercise as medicine" for adolescents with bipolar disorder (BD). Numerous review articles attest to widespread recognition that aerobic exercise (AE) could be an important part of the treatment armamentarium to reduce the symptom burden, neurocognitive dysfunction, and cardiovascular disease (CVD) risk, improve quality of life (QOL), and even engage core biological treatment targets in BD. It appears self-evident that treatment for adolescents with BD, who experience high symptom burden, neurocognitive deficits, and increased CVD risk, should target their aerobic fitness (AF), yet there is not a single study in the world literature on this topic. Remarkably, there have been no intervention studies that specifically focus on aerobic exercise or that directly evaluate changes in AF in any BD age group. Overall physical activity is important, but focusing on AF offers unique potential benefits in terms of simultaneously ameliorating and enhancing mood, neurocognition, and cardiovascular health. Importantly, a recent American Heart Association (AHA) Scientific Statement confirms that it is the most aerobically unfit for whom even modest improvements in AF offer the greatest relative benefits. Nonetheless, important questions arise as to whether and how AF in this population can be improved. There is a clear and unmet need for effective behavior change counseling (BCC) interventions targeting AF that are tailored to the unique needs of adolescents with BD.

DETAILED DESCRIPTION:
The overarching goal of this project is to advance the field in terms of BCC approaches to improving AF among adolescents with BD, a group for whom improvements in AF offer multiple parallel benefits. This project will serve as a preliminary feasibility study, a necessary step in the path toward a well-powered, randomized controlled trial (RCT). If exercise is to achieve the same status as other evidence-based treatments for adolescents with BD, it will be necessary to evaluate exercise with the same level of rigor as other interventions. A crucial first step toward the ultimate goal of an adequately powered RCT is to demonstrate that adolescents with BD will enroll in, and actively participate in, an intervention study that accurately reflects what would be required of participants in such a study.

Objective 1: Evaluate the feasibility of developing a 24-week BCC intervention, customized and personalized for adolescents with BD, focusing on increasing AF.

Objective 2: Evaluate the feasibility of implementing the 24-week BCC intervention.

Objective 3: Evaluate the feasibility of measuring the effects of the intervention.

Exploratory: Examine the impact on AF of a 24-week BCC intervention, customized and personalized for adolescents with BD. Related hypothesis-generating analyses will examine the impact of specific variables (e.g., mood, medications, exercise-induced feelings, specific BCC modules, changes in motivation and self-efficacy) on AF changes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 13-21 years old
* Meet diagnostic criteria for BD (using KSADS-PL)
* Report moderate-vigorous exercise <150 minutes/week in the preceding 12 weeks
* Written clearance from primary care physician required

Exclusion Criteria:

* Unable to provide informed consent (e.g., severe psychosis, IQ<80)
* Presence of hypo/hypertension and history of exercise induced and aggravated conditions that are contraindications to proceeding with the study (e.g., syncope, asthma)
* Known cardiac condition (e.g., conduction abnormality, congenital heart disease) or other active medical condition that precludes aerobic exercise
* Known respiratory condition that precludes aerobic exercise
* Known health condition of physiological impairment that would preclude participation in exercise
* Currently manic (PSR score of 5 or 6 on mania)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Barriers to participation using the Client Satisfaction Questionnaire | Week 12
Barriers to participation using the Client Satisfaction Questionnaire | Week 24
Satisfaction of patient, parent, and consumer advocate co-investigators using the Client Satisfaction Questionnaire | Week 12
Satisfaction of patient, parent, and consumer advocate co-investigators using the Client Satisfaction Questionnaire | Week 24
Percentage of target sample size enrolled | three years (At the end of study completion)
Percentage of screened participants meeting inclusion criteria comparing number of participants screened to number of participants who meet inclusion criteria | Three years
  Evaluating whether sample reflects clinical population in which exercise is an anticipated intervention
Barriers to recruitment | Three years
  Qualitative assessment using phenomenological approach
Therapist adherence with behavior change counseling using the Behavior Change Counseling Index | three years
Participant attendance | Week 0
  Attendance at core sessions
Participant attendance | Week 4
  Attendance at core sessions
Participant attendance | Week 8
  Attendance at core sessions
Participant attendance | Week 12
  Attendance at core sessions
Participant attendance | Week 1
  Attendance at phone calls/texting sessions
Participant attendance | Week 2
  Attendance at phone calls/texting sessions
Participant attendance | Week 3
  Attendance at phone calls/texting sessions
Participant attendance | Week 5
  Attendance at phone calls/texting sessions
Participant attendance | Week 6
  Attendance at phone calls/texting sessions
Participant attendance | Week 7
  Attendance at phone calls/texting sessions
Participant attendance | Week 9
  Attendance at phone calls/texting sessions
Participant attendance | Week 10
  Attendance at phone calls/texting sessions
Participant attendance | Week 11
  Attendance at phone calls/texting sessions
Participant attendance | Week 16
  Attendance at phone calls/texting sessions
Participant attendance | Week 20
  Attendance at phone calls/texting sessions
Participant completion of daily activity logs | three years
  Number of daily activity logs completed for each participant
Participant attendance | Week 1
  Attendance at exercise coaching session
Percentage of participants who selected the exercise coaching optional module | three years
Percentage of participants who selected the family focused counseling optional module | three years
Percentage of participants who selected the peer support optional module | three years
Percentage of participants who completed the 24 weeks of the study | three years
Percentage of participants who completed the 12 week intervention | three years
Percentage of participants who completed all aerobic fitness testing sessions | three years
Percentage of sessions attended by each team member | three years

SECONDARY OUTCOMES:
Change in aerobic fitness using the Modified Bruce Protocol | From week 0 to week 12
  The modified Bruce Treadmill Test (weeks 0, 12) progresses through stages every 3 minutes, with each stage increasing in incline of the treadmill platform and increasing speed of treadmill belt. The modified Bruce treadmill test will provide an estimation of VO2max based on treadmill time.
Change in aerobic fitness using the Modified Bruce Protocol | From week 12 to week 24
  The modified Bruce Treadmill Test (weeks 12, 24) progresses through stages every 3 minutes, with each stage increasing in incline of the treadmill platform and increasing speed of treadmill belt. The modified Bruce treadmill test will provide an estimation of VO2max based on treadmill time.
Change in aerobic fitness using the Modified Canadian Aerobic Fitness Test | From week 2 to week 8
  The modified Canadian AF Test (weeks 2, 8), consists of stepping up and down two steps (20.3 cm in height each) during 3-minute stages while listening to set cadences. The stepping rate will depend on age and sex, and participants will be required to reach a target heart rate of 85% of predicted maximum (220 - age). VO2 max will be estimated through the following equation: VO2 max = 32.5 +13.6 x estimated oxygen cost (L/min) - 0.24 x age - 0.17 x weight (Kg).
Schedule for Affective Disorders and Schizophrenia for School Age Children, Present and Life Version (K-SADS-PL) | baseline
  The K-SADS-PL is a semi-structured interview designed to ascertain present episode and lifetime history of psychiatric illness, according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria for children and adolescents.
Longitudinal Interval Follow-up Evaluation (LIFE) | baseline, week 12, week 24
  The LIFE will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study
Brief Quality of Life in Bipolar Disorder (QoL.BD) | baseline, week 12, week 24
  The Brief QoL.BD is a self-report that will be used to assess condition-specific quality of life. Scale responses include: strongly disagree, disagree, neutral, agree, and strongly agree. The scale assesses 12 basic domains of quality of life: physical, sleep, mood, cognition, leisure, social, spirituality, finances, household, self-esteem, independence, and identity. Total scores can range from 12-60 with 60 identifying a high quality of life.
36-Item Short Form Health Survey (SF-36) | baseline, week 12, week 24
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. To score, first, precoded numeric values are recoded per the scoring key given (see link). Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Table 2 lists the items averaged together to create each scale. Items that are left blank (missing data) are not taken into account when calculating. https://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html
Client Satisfaction Questionnaire-8 (CSQ-8) | At weeks 12 and 24
  The Client Satisfaction Questionnaire-8 will be used to assess intervention satisfaction. An overall score is calculated by summing the respondent's rating (item rating) score for each scale item. For the CSQ-8 version, scores therefore range from 8 to 32, with higher values indicating higher satisfaction. Scoring values range from 1-4 with 4 meaning high satisfaction and 1 meaning low satisfaction.
The Stages of Change Questionnaire (SCQ) | baseline, week 4, week 8, week 12, and week 24
  The Stages of Change Questionnaire is a self-report that will provide the stage of behavior change relating to exercise status for discussion at BCC sessions. Six statements are provided and the participant is asked to select the statement that best describes them. This will then determine which stage of change they are in (precontemplation, contemplation, preparation, action, maintenance, or relapse).
Outcome Expectations for Exercise (OEE) | baseline, week 12, week 24
  The Outcome Expectations for Exercise tool will assess expectations of the benefits from physical activity. The Outcome Expectations for Exercise Scale contains 9 statements rated by participants using a 5-point likert scale from 1 "Strongly Disagree" to 5 "Strongly Agree". If negative or low expectations are found, an intervention can be implemented that may increase the expectancy of exercise and therefore create a more active lifestyle.
Motives for Physical Activities Measure-Revised (MPAM-R) | baseline, week 12, week 24
  The MPAM-R will assess motives for activity participation. There are five categories: interest/enjoyment, competence, appearance, fitness, and social. It is rated on a likert scale ranging from 1 (not at all true for me) to 7 (very true for me).
Behavioral Regulation in Exercise Questionnaire (BREQ-3) | baseline, week 12, week 24
  The Behavioral Regulation in Exercise Questionnaire-3 is a 24-item self-report scale that assesses the reasons why people exercise. Questions range from 0 (not true for me) to 4 (very true for me). BREQ has been used either as a multidimensional instrument giving separate scores for each subscale, or as a unidimensional index of the degree of self-determination, known as the relative autonomy index. In order to use the BREQ as multidimensional scales, the mean scores are calculated for each set of items into categories (amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic regulation).
Exercise Self-Efficacy | baseline, week 12, week 24
  This measure will assess exercise-related self-efficacy. An 11-point scale is used with 1 indicating "not at all confident" and 7 indicating "very confident". Participants can also endorse 0 "does not apply to me". High scores indicate high levels of self-efficacy.
Quick Weight, Activity, Variety, and Excess Screener (WAVE) | baseline, week 12, week 24
  WAVE is a 17-item self-report instrument that ascertains 5 subscales: weight, physical activity, dietary variety, dietary excess, and household food insecurity. The scores for each question can be added to generate an overall WAVE score that provides a quick estimate of the patient's overall health habits. The WAVE score can range from 0 to 21. The scores are interpreted as follows: 0 to 5= High priority for intervention to improve health habits; 6 to 11=In need of much improvement; 12 to 16=Some good health habits but needs improvement; and 17 to 21=Good to excellent health habits.
Drug Use Screening Inventory (DUSI) | baseline, week 12, week 24
  Assesses drug use
Stressful Life Events Schedule (SLES) | baseline, week 12, week 24
  The SLES (total score) ascertains 80 adolescent- and parent-reported negative life events, and their impact, during the preceding six months or time since last assessment. Participants responds whether or not an event has occurred and then rate how much the event affected them on a scale of 1 to 4 (1=not at all to 4=a lot).
Pittsburgh Sleep Quality Index (PSQI) | baseline, week 12, week 24
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month time interval. Each question is scored with a total score of "5" or greater indicating poor sleep quality. Items collect time and length of sleep. Other items look at factors affecting sleep and responses range from 0 (not during the past month) to 3 (three or more times a week).
Exercise-Induced Feeling Inventory (EIFI) | baseline, then pre- and post-aerobic fitness testing at weeks 0, 2, 8, 12, and 24
  The Exercise-Induced Feeling Inventory measures the intensity of 12 feeling states as they occur in relation to physical activity. Responses are rated from 0 (do not feel) to 4 (feel very strongly) for each emotion. The EIFI consists of 12 items that capture 4 distinct feeling states: revitalization, tranquility, positive engagement, and physical exhaustion. The EIFI consists of 4 distinct subscales. Subscale scores are obtained by summing or averaging the numerical values chosen for the adjectives within a particular subscale. The four subscales include: (1) Positive Engagement (items 4, 7, & 12), (2) Revitalization (items, 1, 6, & 9), (3) Tranquility (items 2, 5, & 10), and (4) Physical Exhaustion (items, 3, 8, & 11).
Physical Activity Logs | Through study completion, an average of 24 weeks
  The physical activity logs will be used by participants to record any moderate to vigorous intensity exercise, including details such as the time of day, type of exercise, and thoughts, feelings and physical sensations in regards to the exercise

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, PhD, Principal Investigator — Senior Scientist, Psychiatrist
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No